CLINICAL TRIAL: NCT06481982
Title: Value of Advanced MRI Techniques in the Assessment of Endometriosis
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Advanced MRI Endometriosis
Record Dates: First submitted 2024-06-19; First posted 2024-07-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI sequences

SUMMARY:
Endometriosis is a common gynaecological disease, mostly in women of reproductive age, with a prevalence of about 10 %, which is defined by the presence of endometrial-type tissue outside the uterine cavity. Endometriosis is usually limited to the abdominal and especially the pelvic cavity, extra-abdominal lesions are rare. Within the pelvis it shows a wide variety of locations predominantly affecting the ovaries and the uterus or the peritoneum, uterine ligaments and other pelvic structures. Traditionally, there are three major phenotypes of endometriosis: Ovarian endometrioma (OMA), superficial peritoneal endometriosis (SPE), and deep infiltrating endometriosis (DIE). A lesion is considered a DIE, if it shows infiltration deeper than 5 mm into the peritoneum. The ectopic endometrial implants may induce inflammatory processes, causing scar tissue formation, adhesions, and consequently pelvic anatomy distortion.

The prospective study aims to investigate the value of advanced MRI techniques to improve the assessment of pelvic endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo clinically indicated MR imaging for endometriosis evaluation.

Exclusion Criteria:

* Non-MRI compatible devices/implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing routine MRI for endometriosis staging.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 5 years
  Diagnostic accuracy of different MRI sequences in comparison to ultrasound assessment and/or laparoscopy as standard of reference.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided